CLINICAL TRIAL: NCT00079404
Title: A Phase I Study of 17-AAG in Relapsed/Refractory Pediatric Patients With Solid Tumors or Leukemia
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Young Patients With Relapsed or Refractory Solid Tumors or Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01811; ADVL0316; CDR0000355714; COG-ADVL0316; U01CA097452 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Acute Undifferentiated Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tanespimycin

ARMS (1):
- Arm I (Experimental): Patients with solid tumors receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 60-120 minutes on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin in treating young patients with relapsed or refractory solid tumors or leukemia. Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and recommended phase II dose of 17-AAG administered as a 60 or 120-minute intravenous infusion on days 1, 4, 8, and 11, of a 21-day course, to children with refractory solid tumors or relapsed leukemia.

II. To define and describe the toxicities of 17-AAG administered on this schedule.

III. To characterize the pharmacokinetics of 17-AAG in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of 17-AAG within the confines of a phase I study.

II. To assess the biologic activity of 17-AAG. III. To examine the role of CYP3A5 polymorphisms in the pharmacologic and clinical phenotypes observed following administration of 17-AAG to children, within the confines of a phase 1 study.

OUTLINE: This is a dose-escalation, multicenter study.

Patients with solid tumors receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 60-120 minutes on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 6 additional patients with leukemia receive 17-AAG at the MTD as above. If these 6 patients tolerate this regimen, another 6 leukemia patients receive 17-AAG IV over 60 minutes on days 1, 4, 8, 11, 15, and 18.

Treatment repeats every 28 days for 17 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of solid tumor or leukemia with documented M3 marrow

  * Histologic confirmation of intrinsic brain stem tumors not required
* Relapsed or refractory disease
* No known curative therapy
* In patients with CNS tumors, neurologic deficits must be stable for at least the past week
* Performance status - Karnofsky 50-100% (>10 years of age)
* Performance status - Lansky 50-100% (≤ 10 years of age)
* For patients with solid tumors:

  * Absolute neutrophil count ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3 (transfusion independent)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
* For patients with leukemia:

  * Platelet count ≥ 20,000/mm^3 (may receive platelet transfusions)
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine clearance OR radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine based on age as follows:

  * ≤ 0.8 mg/dL if ≤ 5 years of age
  * ≤ 1.0 mg/dL if > 5 years and ≤ 10 years of age
  * ≤ 1.2 mg/dL if > 10 years and ≤ 15 years of age
  * ≤ 1.5 mg/dL if > 15 years and ≤ 21 years of age
* No uncontrolled infection
* No prior severe allergy to eggs
* No situation that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 7 days (or window for adverse effects has passed) since prior biologic therapy and recovered
* At least 7 days since prior hematopoietic growth factors
* At least 2 months since prior stem cell transplantation and no evidence of graft-vs-host disease
* No concurrent hematopoietic growth factors
* No concurrent biologic therapy
* No concurrent immunotherapy
* At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas) and recovered
* No other concurrent chemotherapy
* No concurrent steroid therapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 3 months since prior total body irradiation or craniospinal radiotherapy
* At least 3 months since prior radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since prior substantial bone marrow radiotherapy
* Recovered from prior radiotherapy
* No concurrent radiotherapy
* No other concurrent investigational drugs
* No other concurrent anticancer agents
* No concurrent phenytoin or phenobarbital
* No concurrent warfarin

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2004-03; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
MTD defined as the maximum dose at which fewer than one-third of patients experience DLT | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Weigel, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States